CLINICAL TRIAL: NCT04537559
Title: Impact of the COVID-19 Pandemic on the Morbidity and Mortality of Non-COVID-19 Patients Hospitalized Around the Epidemic Peak in the Geneva Area (Switzerland) (No COVID Impact)
Brief Title: Impact of COVID-19 Outbreak on Non-COVID-19 Patients
Acronym: NoCOVImpact
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Geneva (Other)
Collaborators: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Jerome Stirnemann, Dr, University Hospital, Geneva
Other Study IDs: 2020-01017
Record Dates: First submitted 2020-08-27; First posted 2020-09-03 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: COVID-19 Outbreak; non COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pre-COVID-19 period: Patients hospitalized between 1.3.2019 and 28.02.2020
- per-COVID-19 period: Patients hospitalized between 1.3.2020 and 28.02.2022
- post-COVID-19 period: Patients hospitalized between 1.3.2022 and 28.02.2023

SUMMARY:
The Geneva Canton organized the health crisis of the COVID-19 epidemic around the care of COVID patients at the University Hospital (HUG), by moving the care of non-COVID patients to private hospitals of the canton. The COVID epidemic appears to have been associated with a decrease in consultations and care for non-COVID patients. An excess of morbidity and mortality (non-COVID) would be possible during or after the epidemic in connection with this "under-medicalization" of non-COVID patients.

The aim of this study is to measure and analyze the impact on the morbidity and mortality of inpatients during and after the COVID-19 epidemic in the adult inpatient wards of HUG and township hospitals / clinics.

DETAILED DESCRIPTION:
The analysis of the various results will be carried out on all HUGs and on the various hospitals / clinics in the canton.

A survival analysis for the outcome of death or rehospitalization will be performed, with a comparison according to each period.

After epidemy evolution, finally, the outcomes will be compared between periods pre-COVID (from 01 march 2019 to 28 february 2020) versus per-COVID (01 march 2020 to 28 february 2022), and versus post-COVID (01 march 2022 to 28 february 2023). And comparaison would be performed between periods during the wave (per-wave) versus periods inter-wave.

A description will be made in number (%) for numerical data and in median (IQR) for quantitative data. Univariate comparisons between the different periods will be carried out by statistical tests, parametric or not, adapted according to the data (Chi2 or Fisher's test for qualitative data, Student's test or Mann-Whitney-Wilcoxon for quantitative data). Statistical significance will be retained in the event of p <0.05.

Multivariate analysis will be performed by logistic regression for the main outcome and by cox model for survival analysis. Different variables will be included in the models, including data on gender, age and comorbidity, as well as any variable having a difference with p <0.2 in univariate analysis.

Secondary analyzes will be carried out by pathology (as the main diagnosis) according to the specific results defined for each situation. In retrospective analysis, these specific data will be relatively limited on the HUG area of full analysis brings together around total of 240,000 hospital stays. The main outcome data will be complete with no missing data. On the other hand, since this is retrospective data, it is possible that some important variables are missing. In this case, other patient data with missing data will not be included in the multivariate analyzes. In the event of missing data greater than 10%, a second sensitivity analysis may be performed after replacing the missing data with a multiple imputation method.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in an adult department
* During the pre-period-COVID-19 period, the per-COVID-19 or the post-COVID-19 periods ie from the 1st march 2019 to 28 february 2023.

Exclusion Criteria:

* Patients who have been hospitalized for COVID-19 infection
* Patients hospitalized in the Department of Adolescent Woman and Child, Department of Psychiatry or Intensive Care Department during the same periods.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized in Geneva hospital or clinic from the 1st march 2019 to 28 february 2023.
Sampling Method: Non-Probability Sample
Enrollment: 240000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Intra-hospital mortality | Assessed at the discharge date, up to 3 months after admission
  death during hospitalization of each patient
composite outcome (worsening during hospitalization) | At the discharge date of hospitalization, up to 3 months after admission
  intra-hospital mortality and / or transfer to intensive care and / or transfer to intermediate care during hospitalization

SECONDARY OUTCOMES:
Pathologies leading to hospitalization | At the discharge date of hospitalization, up to 3 months after admission
  Primary and secondary diagnosis during hospitalization (CIM10 codes)
overall mortality at 3 months (90 days) | within the 3 months after the admission date
  intra or extra hospital mortality : death occuring during hospitalization or after
Potentially avoidable readmission rate | During the 30 days after the patient's discharge
  Potentially avoidable readmission according to SQLape algorithm (http://www.sqlape.com/READMISSIONS.htm)
mortality rate by pathology at 3 months | within the 3 months after the admission date
  mortality for each top 10 of pathologies (intra or extra hospital mortality for each pathology)
length of stay | At the discharge date of hospitalization, up to 3 months after admission
  Hospital length of stay (Time between admission date and discharge date)
rate of transfer to intermediate or intensive care | At the discharge date, up to 3 months after admission
  Number of patients with transfer to intensive or intermediate care during hospitalization
rate of transfer to rehabilitation care | At the discharge date of acute care, up to 3 months after admission
  Number of patients with rehabilitation transfer during hospitalization
specific gravity outcomes for patients with pneumonia : CURB 65 scale (Confusion, Urea, Respiratory rate, Blood pressure, Age [>65]) | At the acute care admission
  CURB65 scale: min-max 0 to 5 points [5 points : worse outcome]
specific gravity outcomes for patients with cardiac Failure : KILLIP class | At the acute care admission
  KILLIP class (class 1 to 4) [class 4 : worse outcome]. The KILLIP classification is a system used in individuals with an acute myocardial infarction (heart attack), taking into account physical examination and the development of heart failure in order to predict and stratify their risk of mortality.
specific gravity outcomes for patients with cardiac Failure : Weight variation | At the acute care admission
  Weight variation : variation of weight at the admission compared to the basis weight
specific gravity outcomes for patients with cardiac Failure or lung disease | At the acute care admission
  FIO2 (% O2 prescribed): Fraction of inspired oxygen
Leukocytes serum level | At the acute care admission
  Giga / litre
Polynuclear neutrophils serum level | At the acute care admission
  Giga / litre
Lymphocytes serum level | At the acute care admission
  Giga / litre
Hemoglobin serum level | At the acute care admission
  gram/litre
Thrombocytes serum level | At the acute care admission
  Giga / litre
Quick serum level | At the acute care admission
  in %
INR (International Normalized Ratio) | At the acute care admission
  No unit
fibrinogen serum level | At the acute care admission
  gram/litre
PTT serum level (partial Thromboplastin time) | At the acute care admission
  in second
D-Dimers serum level | At the acute care admission
  ng / ml
glucose serum level | At the acute care admission
  mmol / litre
glycated hemoglobin serum level (HbA1C) | At the acute care admission
  in %
C-reactive protein serum level (CRP) | At the acute care admission
  mg / litre
sodium serum level | At the acute care admission
  mmol / l
potassium serum level | At the acute care admission
  mmol / l
chlorides serum level | At the acute care admission
  mmol / l
calculated osmolality serum level | At the acute care admission
  mOsm / kg
Phosphates serum level | At the acute care admission
  mmol / l
corrected calcium serum level | At the acute care admission
  mmol / l
urea serum level | At the acute care admission
  mmol / l
creatinine serum level | At the acute care admission
  µmol / l
eGFR (CKD-EPI) serum level | At the acute care admission
  ml / min / 1.73m2
albumin serum level | At the acute care admission
  g / l
prealbumin serum level | At the acute care admission
  mg / l
cyanocobalamin serum level | At the acute care admission
  pmol / l
folate serum level | At the acute care admission
  nmol / l
25-hydroxy vitamin D (D2 + D3) serum level | At the acute care admission
  nmol / l
proBNP (Brain Natriuretic Peptid) serum level | At the acute care admission
  ng / l
Ultra sensitive Troponin T serum level | At the acute care admission
  ng / l
ASAT (aspartate transaminase) serum level | At the acute care admission
  U / l
ALAT (alanine aminotransferase) serum level | At the acute care admission
  U / l
Alkaline phosphatases serum level | At the acute care admission
  U / l
Gamma glutamyl transpeptidase. serum level | At the acute care admission
  U / l
Total bilirubin serum level | At the acute care admission
  µmol / l
ferritin serum level | At the acute care admission
  µg / l
TSH serum level | At the acute care admission
  mU / l
Arterial pH | At the acute care admission
  No unit
Arterial pCO2 (carbon dioxide partial pressure) | At the acute care admission
  kPa
Arterial pO2 (oxygen partial pressure) | At the acute care admission
  kPa
Arterial lactate | At the acute care admission
  mmol / l
Arterial HCO3 (bicarbonate) | At the acute care admission
  mmol / l
protein serum level | At the acute care admission
  g / l
Arterial pressure | At the acute care admission
  Arterial pression (min-max), in mmHg
cardiac rates | At the acute care admission
  Bat/mn
respiratory rates | At the acute care admission
  /mn
temperature | At the acute care admission
  Celsius degrees
oxygen saturation | At the acute care admission
  Percutaneous oxygen saturation (in %)
peak flow | At the acute care admission
  L/mn
specific scales : VAS of pain | At the acute care admission
  Visual analog Pain scale (min-max : 1 to 10 [worse outcome])
specific scales : FIM | At the acute care admission
  Functional Independence Measure (min-max : 18 [worse outcome]) to 126)
specific scales : SOFA score | At the acute care admission
  Sequential Organ Failure Assessment Score (min-max : 0 to 24 [worse outcome])
specific scales : MNA | At the acute care admission
  Mini Nutritional Assessment (min-max : 0 [worse outcome] to 14)
specific scales : NRS | At the acute care admission
  Nutrition Risk Screening (min-max : 0 to 12 [worse outcome])
serum or urine positive bacteriologic sample | At the acute care admission or during hospitalization
  number of positive hemoculture or urinary cultures
Patient questionnaire | At the discharge date of hospitalization, up to 3 months after admission
  Questionnaire asking each patient if they had difficulty seeing a doctor before their hospitalization and if they delayed their hospitalization due to the COVID-19 crisis.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Stirnemann, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welt FGP, Shah PB, Aronow HD, Bortnick AE, Henry TD, Sherwood MW, Young MN, Davidson LJ, Kadavath S, Mahmud E, Kirtane AJ; American College of Cardiology's Interventional Council and the Society for Cardiovascular Angiography and Interventions. Catheterization Laboratory Considerations During the Coronavirus (COVID-19) Pandemic: From the ACC's Interventional Council and SCAI. J Am Coll Cardiol. 2020 May 12;75(18):2372-2375. doi: 10.1016/j.jacc.2020.03.021. Epub 2020 Mar 19. No abstract available. PMID 32199938
- [Background] Garcia S, Albaghdadi MS, Meraj PM, Schmidt C, Garberich R, Jaffer FA, Dixon S, Rade JJ, Tannenbaum M, Chambers J, Huang PP, Henry TD. Reduction in ST-Segment Elevation Cardiac Catheterization Laboratory Activations in the United States During COVID-19 Pandemic. J Am Coll Cardiol. 2020 Jun 9;75(22):2871-2872. doi: 10.1016/j.jacc.2020.04.011. Epub 2020 Apr 10. No abstract available. PMID 32283124
- [Background] Roffi M, Guagliumi G, Ibanez B. The Obstacle Course of Reperfusion for ST-Segment-Elevation Myocardial Infarction in the COVID-19 Pandemic. Circulation. 2020 Jun 16;141(24):1951-1953. doi: 10.1161/CIRCULATIONAHA.120.047523. Epub 2020 Apr 21. No abstract available. PMID 32315205
- [Background] Rosenbaum L. The Untold Toll - The Pandemic's Effects on Patients without Covid-19. N Engl J Med. 2020 Jun 11;382(24):2368-2371. doi: 10.1056/NEJMms2009984. Epub 2020 Apr 17. No abstract available. PMID 32302076
- [Background] Killip T 3rd, Kimball JT. Treatment of myocardial infarction in a coronary care unit. A two year experience with 250 patients. Am J Cardiol. 1967 Oct;20(4):457-64. doi: 10.1016/0002-9149(67)90023-9. No abstract available. PMID 6059183